CLINICAL TRIAL: NCT07363135
Title: Evaluation of Albumin Platelet-Rich Fibrin Application Following Scaling and Root Planing on Gingival Crevicular Fluid Growth Factors in Patients With Periodontitis
Brief Title: Evaluation of Albumin Platelet-Rich Fibrin Following SRP in Patients With Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/248A
Record Dates: First submitted 2025-12-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Periodontitis; Periodontitis (Stage 3)
Keywords: periodontitis; prf; platelet rich-fibrin; Non-surgical periodontal treatment; Albumin prf; platelet-derived growth factor; vascular endothelial growth factor; basic fibroblast growth factor; transforming growth factor-beta
MeSH Terms: conditions — Periodontitis; Camurati-Engelmann Syndrome

STUDY DESIGN:
Intervention Model Description: This study utilized a split-mouth, within-subject design rather than a classical crossover or parallel group design. Each subject received both the intervention (Alb-PRF) and control (no Alb-PRF) on different sites of the oral cavity.
Who Masked: Participant
Masking Description: In addition to masking the participants, the researcher who performed the biochemical analyses was also masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Site (Experimental): Application of Alb-PRF to periodontal pockets in the test sites.
  Interventions: Procedure: Albumin platelet-rich fibrin
- Control Site (Sham Comparator): Control sites received a sham intervention consisting of sterile saline solution irrigation into the periodontal pockets, to mimic the procedural aspects of PRF placement without delivering any biologically active material.
  Interventions: Other: Sterile saline (0.9%)

INTERVENTIONS:
Procedure: Albumin platelet-rich fibrin — Application of Alb-PRF to the periodontal pockets in the test sites.
  Arms: Test Site
Other: Sterile saline (0.9%) — Control sites received a sham intervention consisting of sterile saline solution irrigation into the periodontal pockets, to mimic the procedural aspects of PRF placement without delivering any biologically active material.
  Arms: Control Site

SUMMARY:
The study aims to investigate whether application of albumin platelet-rich fibrin (Alb-PRF) into the gum pockets after scaling and root planing (SRP) can improve healing in patients with Stage III Grade B periodontitis. Periodontitis is a chronic disease that damages the tissues and bone surrounding the teeth and can lead to tooth loosening or loss if untreated. SRP is the first and most important treatment step, cleaning the tooth surfaces and smoothing the roots to reduce inflammation, but healing is often limited. PRF, made from the patient's own blood, is rich in platelets and growth factors that support tissue repair, and Alb-PRF is a new form that stays longer in the pocket and releases growth factors over time. In this study, 23 patients who meet the inclusion criteria (adults without systemic diseases, not using medications, non-smokers, not pregnant or breastfeeding, and not recently treated for periodontitis) will participate in a split-mouth design, where one side of the mouth receives SRP+ Alb-PRF and the other side receives SRP alone. Clinical measurements, including plaque, gum inflammation, bleeding, pocket depth, gum recession, and attachment levels, will be taken at baseline, 3 months, and 6 months, while X-rays will assess bone defects at baseline and 6 months. Additionally, gingival crevicular fluid (GCF) will be collected from the deepest pockets at baseline and on days 7, 14, and 21 to measure growth factors in the laboratory. Blood from patients will be processed to prepare the albumin-PRF gel, which will be carefully applied to the deep pockets on the test side. The investigators expect that pockets treated with albumin-PRF gel will show greater clinical attachment gain and higher, longer-lasting growth factor levels, potentially leading to improved gum and bone healing compared to SRP alone.

DETAILED DESCRIPTION:
The study aims to investigate the effects of applying albumin platelet-rich fibrin (Alb-PRF) into periodontal pockets following scaling and root planing (SRP) on clinical, radiographic, and gingival crevicular fluid (GCF) growth factor parameters in patients with periodontitis. Periodontitis is a chronic inflammatory disease that affects the periodontal ligament and alveolar bone surrounding the teeth, leading to tooth mobility and potential tooth loss if left untreated. SRP represents the initial and most important therapeutic intervention, involving mechanical removal of plaque and calculus, as well as smoothing of root surfaces to reduce inflammation and facilitate healing. While SRP alone can decrease pocket depth and provide some clinical attachment gain, healing is often limited, generally resulting in repair through long junctional epithelium rather than true regeneration. To enhance clinical outcomes and accelerate regeneration, various adjunctive therapies, including local antibiotics, regenerative materials, photodynamic therapy, and laser treatments, have been explored and reported to provide positive effects. In recent years, autologous PRF applied into the periodontal pocket has demonstrated beneficial contributions to both clinical and biochemical parameters, as it is rich in concentrated platelets and alpha granules containing growth factors such as platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), and transforming growth factor-beta (TGF-β), which collectively promote cellular proliferation, differentiation, migration, and wound healing. PRF not only delivers these growth factors but also provides a fibrin matrix that acts as a scaffold to support tissue repair. However, the clinical efficacy of PRF is limited by its relatively short duration in the tissue, with effects diminishing approximately 10 days after application, and absorption occurring within a short time frame. To overcome these limitations, a modified approach has been developed in which the upper plasma fraction (platelet poor plasma, PPP) is heat-treated and mixed with the middle PRF layer to produce an Alb-PRF. This material demonstrates prolonged residence in tissue, delayed resorption, and sustained release of growth factors, while also exhibiting improved mechanical properties compared to conventional PRF. In the present study, 23 patients diagnosed with generalized Stage III Grade B periodontitis based on clinical and radiographic examinations will be enrolled. Eligible participants are adults without systemic diseases, not using medications, non-smokers, and not pregnant or breastfeeding, and who have not received periodontal therapy within the past six months. A randomized controlled split-mouth design will be implemented, with one side of the mouth serving as the test site receiving SRP+Alb-PRF, and the contralateral side serving as the control site receiving SRP alone. Clinical periodontal indices, including plaque index, gingival index, bleeding on probing, probing pocket depth, clinical attachment level, and gingival recession, will be recorded at baseline, 3 months, and 6 months. Radiographic assessment of defect depth, percentage of root involvement, and defect angles will be performed at baseline and 6 months. GCF samples will be collected from the deepest pockets at baseline and on days 7, 14, and 21 post-treatment, isolated using periostrips following removal of supragingival plaque, and analyzed for PDGF-BB, VEGF, b-FGF, and TGF-β concentrations using ELISA at the Gülhane Training and Research Hospital Biochemistry Department. Blood for preparation of Alb-PRF will be drawn from the antecubital vein, centrifuged to separate layers, and the upper plasma fraction heated and mixed with injectable PRF using a three-way serum kit to produce the gel, which will then be carefully applied to deep pockets in the test region without overflow. Clinical, radiographic, and biochemical outcomes will be statistically analyzed using SPSS software, employing paired tests such as dependent t-tests, Wilcoxon, and Friedman tests for intra-subject comparisons, with Pearson correlation analysis for continuous variables, and a significance threshold of p<0.05. The sample size of 23 patients (providing 46 test and control sites) was calculated based on previous studies to achieve 95% statistical power. The investigators hypothesized that Alb-PRF application will result in superior clinical attachment gain and prolonged expression of growth factors compared to SRP alone, thus potentially enhancing both soft tissue and alveolar bone regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Stage 3 Grade B periodontitis
* Being between the ages of 18-65
* Vertical bone defects in two quadrants

Exclusion Criteria:

* Smoking
* Having a systemic disease
* Taking any medication
* Being pregnant or breastfeeding
* Having received chemotherapy, radiotherapy or immunosuppressant treatments
* Having received periodontal treatment in the last 6 months•Having used antibiotics in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Probing Pocket Depth (PPD) | Baseline, 3 months, and 6 months
  Change in probing pocket depth (mm) measured at baseline, 3 months, and 6 months following treatment.
Change in Clinical Attachment Level (CAL) | Baseline, 3 months, and 6 months
  Change in clinical attachment level (mm) measured at baseline, 3 months, and 6 months following treatment.
Concentration of PDGF-BB in Gingival Crevicular Fluid | Baseline, Day 7, Day 14, Day 21
  PDGF-BB concentration (pg/mL) measured in gingival crevicular fluid at baseline and on days 7, 14, and 21 following treatment.
Concentration of VEGF in Gingival Crevicular Fluid | Baseline, Day 7, Day 14, Day 21
  VEGF concentration (pg/mL) measured in gingival crevicular fluid at baseline and on days 7, 14, and 21 following treatment.
Concentration of b-FGF in Gingival Crevicular Fluid | Baseline, Day 7, Day 14, Day 21
  b-FGF concentration (pg/mL) measured in gingival crevicular fluid at baseline and on days 7, 14, and 21 following treatment
Concentration of TGF-β in Gingival Crevicular Fluid | Baseline, Day 7, Day 14, Day 21
  TGF-β concentration (pg/mL) measured in gingival crevicular fluid at baseline and on days 7, 14, and 21 following treatment.

SECONDARY OUTCOMES:
Change in Plaque Index Score | Baseline, 3 months, and 6 months
  Change in plaque index score assessed at baseline, 3 months, and 6 months following treatment.
Change in Gingival Index Score | Baseline, 3 months, and 6 months
  Change in gingival index score assessed using at baseline, 3 months, and 6 months following treatment.
Change in Bleeding on Probing Percentage (%) | Baseline, 3 months, and 6 months
  Change in bleeding on probing expressed as a percentage of bleeding sites assessed at baseline, 3 months, and 6 months following treatmen
Change in Gingival Recession (mm) | Baseline, 3 months, and 6 months
  Change in gingival recession measured in millimeters from the cemento-enamel junction (CEJ) to the gingival margin at baseline, 3 months, and 6 months following treatment
Change in Radiographic Bone Defect Depth (mm) | Baseline and 6 months
  Change in bone defect depth measured on standardized periapical radiographs as the vertical distance from the cemento-enamel junction (CEJ) to the base of the defect at baseline and 6 months following treatment.
Change in Radiographic Bone Loss Percentage Relative to Root Length (%) | Baseline and 6 months
  Change in radiographic bone loss percentage calculated relative to root length. Root length was defined as the distance from the cemento-enamel junction (CEJ) to the point where a line drawn parallel to the long axis of the tooth intersected a horizontal line passing through the root apex, measured at baseline and 6 months.
Change in Radiographic Bone Defect Angle (degrees, °) | Baseline and 6 months
  Change in the radiographic bone defect angle measured on standardized periapical radiographs at baseline and 6 months following treatment. The defect angle was defined as the angle between a line drawn parallel to the long axis of the tooth and a line connecting the cemento-enamel junction (CEJ) to the base of the bone defect.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Faculty of Dentistry, University of Health Sciences, Ankara, Turkey, Ankara, Keçiören, Turkey (Türkiye)